CLINICAL TRIAL: NCT02673658
Title: Project for Cognitive Advancement in Infants With Neuromotor DisOrders:The CAN-DO Project
Brief Title: Project for Cognitive Advancement in Infants With Neuromotor Disorders
Acronym: CAN-Do
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duquesne University (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4100068712 Project 1
Record Dates: First submitted 2016-01-29; First posted 2016-02-04 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Motor Coordination or Function; Developmental Disorder
Keywords: infant development, early intervention
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motor + problem solving (Active Comparator): This method focuses on spontaneous movement (rather than facilitated movement). Self-initiated, functionally directed movement is emphasized. Intervention includes guidance and cues, which gently call the child's attention to the support surface, and a set-up of the environment for small increments of movement so that the child can solve a movement problem. Passive movements are not used. Each small increment of movement to advance sitting skill or other motor skills is paired with a specific object or toy that challenges a cognitive concept for spatial problem solving. In this approach, the parent will adjust toys and supports to encourage changes of position from sitting, to transitions in and out of sitting to crawling or standing, but will not assist the child physically.
  Interventions: Behavioral: Motor + problem solving
- Body weight support training (Active Comparator): In this approach, infants will be supported physically by their parents to take steps, sit, crawl, or reach, in practice sessions focused simply on the motor skill. Toys or problem solving will not be part of this intervention, but the child will be assisted (lifted by the parent) through movement to improve strength and learn specific movements and new positions. The child will be able to perform as much of the movement as possible, but the parents will initiate the activity if the child does not initiate, and the parent will lift the child passively through the task if the child is unable to move.
  Interventions: Behavioral: body weight support training

INTERVENTIONS:
Behavioral: Motor + problem solving — Developmental motor tasks incorporating cognitive concepts such as object permanence
  Arms: Motor + problem solving
Behavioral: body weight support training — Mobility tasks to change positions or move the body with assistance to initiate movement
  Arms: Body weight support training

SUMMARY:
The purpose of this longitudinal study is to examine the ongoing interaction between the domains of cognitive and motor development in infants with neuromotor disability, and to compare outcomes of two groups of infants receiving two different types of home-based, parent-delivered physical therapy intervention, in order to determine which intervention is more effective in advancing cognitive as well as motor development. Knowledge of the effectiveness of two types of intervention will lead to improved early intervention for children with developmental disabilities, as well as future studies to examine ongoing outcomes.

DETAILED DESCRIPTION:
This longitudinal study will examine the ongoing interaction between the domains of cognitive and motor development in infants with neuromotor disability, as well as compare differences between groups of infants receiving two types of intervention.

The specific aims for this study are:

1. To measure the changes of the head, trunk and pelvis as the primary orienting segments of the body during the achievement of sitting and the transition to crawling in infants with neuromotor disability.
2. Describe the changes in problem-solving and cognitive abilities of infants with neuromotor disability as they transition to stable sitting and then to crawling.
3. Using eye-tracking technology, quantify the evolution of focused attention in infants with neuromotor disability as the motor skills of sitting and the transition to crawling emerge.
4. Compare motor skill, visual attention and cognitive change as sitting and crawling emerge between groups of infants with neuromotor disabilities receiving two different interventions, and determine the effects of distinctly different paradigms: one that focuses simply on building motor skill, and the other that builds motor and cognition together.

This is a longitudinal study, with between group comparisons to determine the effectiveness of the intervention, and within group comparisons to determine change over time. Measures will occur in the home at baseline, at the end of month 1 of intervention, the end of month 2, the end of month 3, and at a 9 month follow-up visit, for a total of 5 measurement times. Each session will take approximately 1 hour each time. Because we want to look at the child's movement and posture, the child should be clothed in either an undergarment or a bathing suit that allows a view of their trunk, legs and arms during the 5 measurement sessions. We will video the child's movement and posture and play doing two standardized infant tests during these measurement sessions. The child will sit on the floor as independently as they can and reach for toys and move through as many developmental postures as they can (crawling, pulling to stand, moving in and out of sitting). The parent will always be next to their child during measurement sessions.

Children will participate in one of the parent-delivered interventions for 3-months after being randomized to one of two groups. Both intervention groups are parent-delivered interventions, with differing goals and differing training. Parents will be trained in one of the following approaches:

Motor-based problem solving approach or the body weight support (BWS) approach.

In both of the above approaches, parents will receive weekly, one-hour sessions at home for updates and training from a physical therapist to advance the program for individual infants. Thus, there will be a total of 12 sessions with a therapist. Each program is individualized because no two infants will have exactly the same skill set. This individualization of programs is standard practice for early intervention. Generally, the suggestions will follow standard developmental guidelines, with sequencing of skills presented in the order of normal development. Both of these approaches are currently used in early intervention for young children with developmental disabilities, but we do not know which is more effective, or if either approach is effective.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a diagnosis of a neuromotor disorder such as cerebral palsy, or a birth history and developmental history indicative of cerebral palsy (prematurity, intraventricular hemorrhage, periventricular leukomalacia) will be selected for this study. The infants will be at Gross Motor Function Classification Scale (GMFCS) levels I, II, or III, because infants at levels IV and V would be unlikely to reach the level of sitting independence to enter the study. Additional behavioral inclusion criteria are: between the ages of 9 months and 3 years at the time of entry into the study; the child should already be independent in prop sitting (sitting with arm support) for at least 1 minute, and be able to lift one arm up in sitting (after being placed in sitting) to reach for a toy placed directly in front of them without losing balance

Exclusion Criteria:

* blindness, dislocated hip, pending orthopedic or neurologic surgery which would interrupt the time period of the intervention, additional diagnosis that affects the neuromuscular system such as spina bifida. A child would not qualify for the study if sitting skills were mature. Mature sitting is operationally defined as: the ability to sit independently without using the arms for support for five minutes or more without falling; reaching for toys using both hands at once without disrupting balance; moving in and out of the sitting position independently.

Ages: 7 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12-15 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure | baseline, 1 month, 2 month, 3 months, up to 9 months post baseline
  Longitudinal Gross Motor Function Measure change measures from baseline to: 1 month, 2 months, 3 months and 9 months post baseline

SECONDARY OUTCOMES:
Visual attention - time to switch between 2 targets, and look time | baseline, 1 month, 2 month, 3 months, up to 9 months post baseline
  Longitudinal eye tracking change measures from baseline to: 1 month, 2 months, 3 months and 9 months post baseline
Early Problem Solving Indicator | baseline, 1 month, 2 month, 3 months, up to 9 months post baseline
  Longitudinal Early Problem Solving Indicator change measures from baseline to:,
  1 month, 2 months, 3 months and 9 months post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Regina T Harbourne, PhD, Principal Investigator — Duquesne University
Locations (1):
- Duquesne University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
No plan to make individual participant data available

REFERENCES:
- [Derived] Harbourne RT, Berger SE. Embodied Cognition in Practice: Exploring Effects of a Motor-Based Problem-Solving Intervention. Phys Ther. 2019 Jun 1;99(6):786-796. doi: 10.1093/ptj/pzz031. PMID 30810750